CLINICAL TRIAL: NCT01877941
Title: Clinical Evaluation of Cardiac Output Estimation Based on Pulse Wave Transit Time
Acronym: esCCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Northern California Institute of Research and Education (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency); Drexel University (Other); Nihon Kohden (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UCSF 12-10139
Record Dates: First submitted 2012-12-05; First posted 2013-06-14 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: cardiac output; pulse oximetry; hemodynamics
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac output monitoring (Active Comparator): Patients undergoing surgery who will have their cardiac output monitored by pulmonary artery catheter (PAC) and endotracheal cardiac output monitoring (ECOM) during surgery and during post-surgical recovery, will also have sensors placed on the arm, finger and leg to calculate pulse wave transit time (PWTT) using the estimated Continuous Cardiac Output system (ecCCO).
  Interventions: Device: Pulmonary Artery Catheter (PAC); Device: Endotracheal Cardiac Output Monitor (ECOM); Device: Estimated Continuous Cardiac Output (esCCO)

INTERVENTIONS:
Device: Pulmonary Artery Catheter (PAC) — A catheter is inserted into the pulmonary artery, through the internal jugular vein; cardiac output is indicated by the speed that a temperature gradient dissipates.
Device: Endotracheal Cardiac Output Monitor (ECOM) — An FDA-approved medical device is inserted into the patient's throat; cardiac output is calculated by measuring how electricity moves through the chest.
Device: Estimated Continuous Cardiac Output (esCCO) — Sensors are placed on the arm, finger and leg to calculate Pulse Wave Transit Time (PWTT); the time it takes for the pulse of the heartbeat to travel through the body.

SUMMARY:
The specific aim of this study is to assess whether a device approved by the FDA to measure pulse oximetry can accurately estimate cardiac output.

DETAILED DESCRIPTION:
We will compare three methods for measuring cardiac output: esCCO, PAC, and ECOM. Cardiac output is an important physiological parameter that must be monitored closely during surgery and during an Intensive Care Unit (ICU) stay. The use of a pulmonary artery catheter (PAC) has been the gold standard for accurate cardiac output (CO) measurement. This method requires a catheter to be inserted into the pulmonary artery and cardiac output is indicated by the speed that a temperature gradient dissipates. While the use of the pulmonary artery catheter is widespread, inserting the pulmonary artery catheter is risky, time consuming and requires a high level of skill. For these reasons, new devices have been developed to measure cardiac output.

A second method typically used is called ECOM (Endotracheal Cardiac Output Monitor). A device is inserted into the patient's throat that calculates cardiac output by measuring how electricity moves through the patient's chest.

The third method, estimated Continuous Cardiac Output (esCCO), uses sensors placed on the patient's finger, arm and chest to calculate Pulse Wave Transit Time (PWTT); the time it takes for the heart beat pulse to travel through the patient's body. The esCCO system is FDA approved for safety and efficacy to measure noninvasive blood pressure and pulse oximetry. The purpose of this study is to assess whether the PSTT calculation provides a cardiac output measure that is comparable to the other methods.

This study is sponsored by Nihon Kohden Corporation who owns and manufactures the esCCO system.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery where cardiac output will be measured with PAC and ECOM.

Exclusion Criteria:

* Failure to obtain consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Wallace, MD, PhD, Principal Investigator — San Francisco Veteran's Admnistration Medical Center
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - Drexel University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cardiac Output Monitoring
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cardiac Output Monitoring
Number analyzed (Participants) | 39
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 65 [55 to 80]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: esCCO (Estimated Continuous Cardiac Output) Monitor
Description: 6 Measurements of cardiac output derived from pulse oximeter measurements using the esCCO system were taken at each time point. The measurements deemed valid under the criteria in the protocol were averaged to represent the reference value at that point. The mean and standard deviation reported consist of the reference values from all time points measured.
  Data for this test were taken at the following timepoints:
  1. Start of Sterenotomy; 2. Before Bypass; 3. 30 Min after bypass; 4. Closure; 5. ICU arrival; 6. 6 hours in ICU; 7. 12 Hours in ICU; 8. 18 Hours in ICU (if PAC still in); 9. 24 Hours in ICU (If PAC still in)
Time Frame: During and after surgery, up to 24 hours
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Cardiac Output Monitoring
Number analyzed (Participants) | 39
liters/minute | 5.6 (1.83)

2. Primary Outcome: PAC (Pulmonary Artery Catheter).
Description: Measurements of cardiac output derived from a PAC (pulmonary artery catheter) using the standard thermodilution technique. At each time point, at least 6 measurements were taken. If, in the opinion of the clinician taking the readings, some of these were in error, more readings were taken to ensure accuracy. In no case were more than 18 readings taken. The points deemed valid by the clinician were averaged to obtain the reference value for that time point. The mean and standard deviation reported consisted of the reference values from all time points measured.
  Data for this test were taken at the following timepoints:
  1. Start of Sterenotomy; 2. Before Bypass; 3. 30 Min after bypass; 4. Closure; 5. ICU arrival; 6. 6 hours in ICU; 7. 12 Hours in ICU; 8. 18 Hours in ICU (if PAC still in); 9. 24 Hours in ICU (If PAC still in)
Time Frame: During and post-surgery, up to 24 hours
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | Cardiac Output Monitoring
Number analyzed (Participants) | 39
liters/minute | 4.95 (1.39)

3. Primary Outcome: Cardiac Output as Measured by ECOM
Description: Measurements of cardiac output derived from the Endotracheal Cardiac Output Monitor (ECOM): An FDA-approved medical device is inserted into the patient's throat; cardiac output is calculated by measuring how electricity moves through the chest.
Time Frame: During and post-surgery, up to 8 hours
Population: Supplies for the ECOM device were not available so it was not tested.
Arm/Group | Cardiac Output Monitoring
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: during surgery and during post-surgical recovery (up to 8 hours)
Groups:
- Cardiac Output Monitoring: Patients undergoing surgery who will have their cardiac output monitored during surgery and during post-surgical recovery. For instance, patients with ischemic heart disease undergoing cardiac bypass graft or percutaneous coronary intervention.
  No adverse events.
Arm/Group | Cardiac Output Monitoring
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No